CLINICAL TRIAL: NCT02760810
Title: Clinical Evaluation of An Approved Contact Lens
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Vision Care, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR-5815
Record Dates: First submitted 2016-05-02; First posted 2016-05-04 (Estimated); Results first posted 2017-07-11 (Actual); Last update posted 2017-07-11 (Actual); Status verified 2017-06

CONDITIONS: Tear Film Characteristics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- narafilcon A (Experimental): Subjects who are new contact lens wearers (neophytes) between the ages of 18-45 will be dispensed the Test Lens and evaluated over a period of 2 weeks.
  Interventions: Device: Marketed Contact Lens

INTERVENTIONS:
Device: Marketed Contact Lens — Narafilcon A

SUMMARY:
This is an 8-visit, bilateral, dispensing clinical study to evaluate the change in tear fluid pH and tear film osmolarity in an FDA-cleared contact lens in new contact lens users over a 14-day period.

ELIGIBILITY:
Inclusion Criteria:

1. The subject must read, understand, and sign the STATEMENT OF INFORMED CONSENT and receive a fully executed copy of the form.
2. The subject must appear able and willing to adhere to the instructions set forth in this clinical protocol.
3. The subject must be between 18 and 45 years of age.
4. The subject must have a valid spectacle prescription with expiration date not over 1 year.
5. The subject's vertex corrected spherical equivalent distance refraction must be in the range of -0.25 Diopters (D) to -6.00 D in each eye.
6. The subject's refractive cylinder must be ≤1.00 Cylindrical Diopter (DC) in each eye.
7. The subject must have best corrected visual acuity of logMAR 0.20 or better in each eye.
8. Subjects should own a wearable pair of spectacles and agree to wear them the day of the initial visit and every morning on subsequent visit days.
9. The subject must be a contact lens neophyte, defined as never having been dispensed contact lenses, or who has taken part in a non-dispensing clinical study or has been fitted with contact lenses in practice but never went on to actually wear the lenses.
10. The subject must have normal eyes (i.e. no ocular medications or infections of any type).

Exclusion Criteria:

1. Currently pregnant or lactating (subjects who become pregnant during the study will be discontinued).
2. Any ocular or systemic allergies or diseases that may interfere with contact lens wear.
3. Any systemic disease, autoimmune disease, or use of medication, which may interfere with contact lens wear.
4. Use of any medication with known tear film effects within 2 weeks prior to and during the study.
5. Entropion, ectropion, extrusions, chalazia, recurrent styes, glaucoma, history of recurrent corneal erosions, aphakia, or moderate or above corneal distortion..
6. Any previous, or planned, ocular or interocular surgery (e.g. radial keratotomy, photorefractive keratectomy (PRK), laser-assisted in situ keratomileusis (LASIK), etc.)
7. Any grade 3 or greater slit lamp findings (e.g. edema, corneal neovascularization, corneal staining, tarsal abnormalities, conjunctival injection) on the FDA classification scale, any previous history or signs of a contact lens-related corneal inflammatory event (e.g. past peripheral ulcer or round peripheral scar), or any other ocular abnormality that may contraindicate contact lens wear.
8. Any ocular infection.
9. Any infectious disease (e.g. hepatitis, tuberculosis) or a contagious immunosuppressive disease (e.g. HIV) by self-report.
10. Any corneal distortion resulting from previous hard or rigid gas permeable contact lens wear.
11. Participation in any contact lens or lens care product clinical trial within 7 days prior to study enrollment.
12. Employee of investigational clinic (e.g. Investigator, Coordinator, Technician).

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2016-04-12 (Actual); Primary Completion 2016-04-26 (Actual); Study Completion 2016-04-26 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Aston University, Birmingham, West Midlands, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 31 subjects were enrolled in this study. Of the enrolled subjects 1 did not meet the eligibility criteria and 30 were dispensed the study lens. Of the dispensed subjects 29 completed the study and 1 subject was discontinued from the study.
Groups:
- Narafilcon A: All subjects wore the same lens throughout the study.
Period: Overall Study
Arm/Group | Narafilcon A
Started | 30
Completed | 29
Not Completed | 1
Not completed — Protocol Violation | 1

BASELINE CHARACTERISTICS:
Population: All subjects that were dispensed a study lens.
Arm/Group | Narafilcon A
Number analyzed (Participants) | 30
Age, Continuous [Mean (Standard Deviation); unit: Years] | 22.8 (4.08)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 11
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian | 18
  White | 12
Region of Enrollment [Number; unit: Participants]
  United Kingdom | 30

OUTCOME MEASURES:

1. Primary Outcome: Tear Film Osmolarity
Description: Tear film osmolarity was measured in each subject eye using the TearLab Osmolarity system. The instrument was placed gently into the lower lid temporal tear minuscus without simulating reflex tearing
Time Frame: 2-Week Follow-up
Population: Subjects that completed all study visits without a major protocol deviation.
Measure: Mean (Standard Deviation); unit: mOsm/L
Units Other Than Participants: Eyes
Arm/Group | Narafilcon A
Number analyzed (Participants) | 27
Number analyzed (Eyes) | 54
mOsm/L | 293.4 (9.50)

2. Secondary Outcome: Tear Film Osmolarity
Description: as for outcome 1
Time Frame: 1-Week Follow-up
Population: Subjects that completed all study visits without a major protocol deviation.
Measure: Mean (Standard Deviation); unit: mOsm/L
Units Other Than Participants: Eyes
Arm/Group | Narafilcon A
Number analyzed (Participants) | 27
Number analyzed (Eyes) | 54
mOsm/L | 294.4 (9.48)

3. Secondary Outcome: Tear Film PH
Description: Tear Film PH was measured using a 1mm Microglass electrode (Thermo Scientific Orion 9810BN) placed gently in lower temporal tear meniscus of non-Schirmer eye without simulating reflex tearing.
Time Frame: 1-Week Follow-up
Population: Subjects that completed all study visits without a major protocol deviation.
Measure: Mean (Standard Deviation); unit: PH value
Arm/Group | Narafilcon A
Number analyzed (Participants) | 27
PH value | 6.86 (0.180)

ADVERSE EVENTS:
Time Frame: Throughout the duration of the study. Approximately 2-weeks per subject.
Arm/Group | Narafilcon A
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days